CLINICAL TRIAL: NCT05074030
Title: Project CHOICE: Developing a Personalized-Feedback EMA/EMI Intervention for Emerging Adults Leaving Psychiatric Partial Hospitalization
Brief Title: EMA/EMI for Psychiatrically Hospitalized Emerging Adults Who Drink to Cope
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2104-001; R34AA028572 (NIH)
Record Dates: First submitted 2021-09-17; First posted 2021-10-12 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNF (Active Comparator): Participants in the PNF condition will receive normative feedback only on their alcohol use.
  Interventions: Behavioral: Personalized Normative Feedback
- PFIcope+EMI (Experimental): The 6-week PFIcope+EMI includes: 1) an in-person personalized feedback session to present feedback on problems with drinking to cope, discuss the individual's use of alcohol to cope, and generate coping skills messages to be used in the EMI intervention; 2) EMA to monitor affect, intention to drink, coping skills usage, alcohol use, drinking to cope post-discharge; 3) tailored text messages (EMI) based on EMA (individualized coping skills messages when NA and intention to drink are reported).
  Interventions: Behavioral: Coping-Motive Specific Personalized Feedback Intervention plus an Ecological Momentary Intervention (PFIcope+EMI)

INTERVENTIONS:
Behavioral: Personalized Normative Feedback — Normative Feedback on drinking behaviors.
  Arms: PNF
Behavioral: Coping-Motive Specific Personalized Feedback Intervention plus an Ecological Momentary Intervention (PFIcope+EMI) — An EMA plus EMI intervention to decrease drinking to cope behaviors among emerging adults receiving psychiatric treatment.
  Arms: PFIcope+EMI

SUMMARY:
The goal of this proposed study is to evaluate an ecological momentary assessment plus an ecological momentary intervention (EMA+EMI) for emerging adults in a psychiatric partial hospitalization program who drink to cope with negative affect (NA) as compared to personalized feedback only. This intervention combines a personalized feedback intervention (PFI) with EMA technology and tailored EMI text messaging (PFICope+EMI). PFICope+EMI not only aims to reduce drinking to cope, but also alcohol use and NA. This study consists of a 6-week randomized controlled treatment trial to test the PFIcope+EMI intervention as compared to personalized normative feedback only (PNF).

DETAILED DESCRIPTION:
Given the relationship between mental health and alcohol problems, there is a need to address comorbidity among emerging adults (EAs) with anxiety and/or depression. The weeks after psychiatric hospitalization are a risky time for problematic alcohol use and recurrence of psychiatric symptoms. The delivery of tailored, coping skills-based, real-time messages could have a significant impact on problematic drinking and depression/anxiety outcomes by reducing the likelihood that an individual drinks to cope with NA.

The aim of this study is to test a 6-week PFIcope+EMI intervention as compared to personalized normative feedback only (PNF) for EA in a partial hospitalization program who drink to cope and binge drink (n=60). The PFIcope+EMI includes: 1) an in-person personalized feedback session to present feedback on problems with drinking to cope, discuss the individual's use of alcohol to cope, and generate coping skills messages to be used in the EMI intervention; 2) EMA to monitor affect, intention to drink, coping skills usage, alcohol use, drinking to cope post-discharge; 3) tailored text messages (EMI) based on EMA (individualized coping skills messages when NA and intention to drink are reported). The Personalized Normative Feedback condition (PNF) will receive a personalized normative feedback report but no EMA or EMI.

Participants' alcohol outcomes and psychiatric symptomatology at 6-weeks, 12-weeks, and 6-months will be assessed to determine outcomes and feasibility/acceptability. It is hypothesized that:

1. Individuals in PFIcope+EMI arm will report between-subjects reductions in drinking to cope, alcohol use, alcohol-related problems, and NA as compared to PNF.
2. PFIcope+EMI will be feasible to implement and result in high rates of participant satisfaction.

Mechanisms that may underlie the efficacy of the intervention for the PFIcope+EMI group utilizing the daily EMA data will be explored. It is hypothesized that:

1. In response to NA, participants will report an increase in coping skills utilization and decreased intent to drink at the following EMA assessment point.
2. NA reductions and increased coping skills utilization will be related to improvements in alcohol use rates and problems at the following EMA assessment.

ELIGIBILITY:
Inclusion Criteria:

1. between 18 and 25 years of age
2. reported alcohol use at least 3x weekly over past month and at least one day per week, on average, of binge drinking (as defined as 4+ drinks/2 hours for men and 3+ drinks/2 hours for women)
3. self-reported use of coping motive (mean of 2+ on coping subscale of MDMQ-R, indicating they drink to cope at least "some of the time")
4. current anxiety and/or depression symptomatology (as assessed CES-D scores above cut-off for high risk for clinical depression and GAD-7 scores above cut-off for moderate to severe anxiety)
5. owns a smartphone capable of downloading EMA app.

Exclusion Criteria:

1. current DSM-5 diagnosis of moderate/severe substance use disorder (other than alcohol, cannabis, or nicotine) as assessed by research staff via SCID
2. a history of psychotic disorder or current psychotic symptoms as assessed by research staff via SCID
3. current suicidal/homicidal ideation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Drinks per Drinking Days | 6-week follow-up
  Drinks per drinking day assessed using the Timeline Followback (TLFB)

SECONDARY OUTCOMES:
Drinking Motives | 6-week follow-up
  Mean Scores on the Drinking to Cope subscale of the Modified Drinking Motives Questionnaire (range from 5 to 25; higher values reflect greater drinking to cope)
Alcohol-related problems | 6-week follow-up
  Number of consequences of alcohol use assessed with the Rutgers Alcohol Problems Index
Alcohol Outcome Expectancies | 6-week follow-up
  The number of benefits and costs associated with changing drinking behaviors as measured by the Alcohol Outcome Expectancies Questionnaire

OTHER OUTCOMES:
Drinks per Drinking Days | 12-week follow-up
  Drinks per drinking day assessed using the Timeline Followback (TLFB)
Drinks per Drinking Days | 6-month follow-up
  Drinks per drinking day assessed using the Timeline Followback (TLFB)
Drinking Motives | 12-week follow-up
  Mean Scores on the Drinking to Cope subscale of the Modified Drinking Motives Questionnaire (range from 5 to 25; higher values reflect greater drinking to cope)
Drinking Motives | 6-month follow-up
  Mean Scores on the Drinking to Cope subscale of the Modified Drinking Motives Questionnaire (range from 5 to 25; higher values reflect greater drinking to cope)
Alcohol-related problems | 12-week follow-up
  Number of consequences of alcohol use assessed with the Rutgers Alcohol Problems Index
Alcohol-related problems | 6-month follow-up
  Number of consequences of alcohol use assessed with the Rutgers Alcohol Problems Index
Alcohol Outcome Expectancies | 12-week follow-up
  The number of benefits and costs associated with changing drinking behaviors as measured by the Alcohol Outcome Expectancies Questionnaire
Alcohol Outcome Expectancies | 6-month follow-up
  The number of benefits and costs associated with changing drinking behaviors as measured by the Alcohol Outcome Expectancies Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Abrantes, Ph.D., Principal Investigator — Butler Hospital/Alpert Medical School of Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No